CLINICAL TRIAL: NCT05940714
Title: Detection of Levels of Periodontopathogens in a Catalan Population of Periodontal Patients Visited in the HOUB
Brief Title: Periodontopathogens of Periodontal Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Barcelona (Other)
Collaborators: Teresa Vinuesa Aumedes (Unknown); Albert Estrugo Devesa (Unknown); Felipe Aguilera Muñoz (Unknown); Ester Fuste Domínguez (Unknown); Enric Jané Salas (Unknown); Isabel Martínez Lizán (Unknown); Sonia Egido Moreno (Unknown); Carlos Omaña Cepeda (Unknown); Alexandra Merlos Gil (Unknown)
Responsible Party: Principal Investigator, José López Lopez, doctor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Perio HOUB
Record Dates: First submitted 2023-06-14; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Periodontal Diseases
Keywords: periodontopathogens; oral hygiene; periodontal patients
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video participants (Experimental): Patients treated at the Hospital Odontològic Universitat de Barcelona (HOUB) who go for a routine visit in the period of the study and wish to participate. Parameters are measured and an oral hygiene teaching intervention is carried out.
  Interventions: Behavioral: Video participants
- Non video participants (No Intervention): Patients treated at the Hospital Odontològic Universitat de Barcelona (HOUB) who go for a routine visit in the period of the study and wish to participate. Parameters are measured and and no initial intervention is performed.

INTERVENTIONS:
Behavioral: Video participants — Showing a video of oral hygiene intructions
  Other Names: Study group
  Arms: Video participants

SUMMARY:
Study the presence of periodontal pathogens in a Catalan population with periodontitis and evaluate the influence of an intervention measure on oral hygiene teaching (video)

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* periodontal disease (grade III and IV)
* gave their informed consent to participate in the study
* do not present associated medical pathology

Exclusion Criteria:

* Patients who do not wish to participate in the study
* Patients following active treatment with antibiotics or having received antibiotic treatment in the last seven days,
* Patients who wear braces.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Presence of periodontopathogens | 1 month
  Study the presence of periodontogens in a Catalan population with periodontitis and evaluate the influence of an intervention measure in the form of oral hygiene education.

SECONDARY OUTCOMES:
Correlate the microbiota and pro-inflammatory cytokine data obtained in the study population with the literature. | 1 month
  Measure through conventional and molecular microbiological study of bacteria, looking for changes in the total count and measurement of cytokine through ELISA/cytometry test and search for quantitative changes
Determine if there are changes in the oral microbiota, before and after an intervention in the form of oral hygiene. | 1 month
  Measure through conventional and molecular microbiological study of bacteria, looking for changes in the total count
Determine if there are changes in the levels of pro-inflammatory cytokines, before and after an intervention measure in the form of oral hygiene. | 1 month
  Measurement through ELISA/cytometry test and search for quantitative changes
Correlate the level of periodontal disease with the patient's oral health. | 1 month
  Classification established in the World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions
Correlate the level of periodontal disease with the patient's systemic diseases | 1 month
  Classification established in the World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions and review of the clinical history
Correlate the variations in the oral microbiota with the patient's systemic diseases. | 1 month
  Measure through conventional and molecular microbiological study of bacteria, looking for changes in the total count and review of the clinical history
Correlate variations in the levels of pro-inflammatory cytokines with the patient's systemic diseases. | 1 month
  Measurement through ELISA/cytometry test and search for quantitative changes and review of the clinical history

CONTACTS AND LOCATIONS:
Locations (1):
- University of Barcelona, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided